CLINICAL TRIAL: NCT05407220
Title: A Randomized, Open-Label, Single-Dose Parallel Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HCP1904 in Healthy Male Volunteers.
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HCP1904 in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-CHORUS-102
Record Dates: First submitted 2022-05-27; First posted 2022-06-07 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group1 (Experimental): Period1: HCP1904-1
  Interventions: Drug: HCP1904-1
- group2 (Experimental): Period1: HCP1904-3
  Interventions: Drug: HCP1904-3

INTERVENTIONS:
Drug: HCP1904-1 — take it once per period
  Arms: group1
Drug: HCP1904-3 — take it once per period
  Arms: group2

SUMMARY:
A Randomized, Open-Label, Single-Dose Parallel Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HCP1904 in Healthy Male Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~45 years in healthy male volunteers
2. Weight ≥ 55kg and BMI 18 ~ 30 kg/m^2
3. Subjects who agree to use medically accepted dual contraceptives up to 14 days after the last administration date of the clinical trial drug and not to provide sperm.
4. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Cmax of Losartan | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
AUC last of Losartan | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
AUC inf of Losartan | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
Tmax of Losartan | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
t1/2 of Losartan | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
CL/F of Losartan | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
Vd/F of Losartan | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
Cmax of EXP3174 | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
AUC last of EXP3174 | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
AUC inf of EXP3174 | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
Tmax of EXP3174 | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
t1/2 of EXP3174 | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
CL/F of EXP3174 | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
Vd/F of EXP3174 | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
Cmax of Chlorthalidone | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
AUC last of Chlorthalidone | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
AUC inf of Chlorthalidone | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
Tmax of Chlorthalidone | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
t1/2 of Chlorthalidone | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
CL/F of Chlorthalidone | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation
Vd/F of Chlorthalidone | Day 1, 2, 3, 4, 5, 7 : pre-dose(0 hour)~144hours
  pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No